CLINICAL TRIAL: NCT04553523
Title: The Hydrus® Microstent New Enrollment Post-Approval Study: A Prospective, Non-Randomized, Multicenter, Single Arm, Clinical Trial
Brief Title: Hydrus® Microstent New Enrollment Post-Approval Study
Acronym: CONFIRM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP 18-001; GLI314-C003 (Other: Alcon Research)
Record Dates: First submitted 2020-09-11; First posted 2020-09-17 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Primary Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Hydrus Microstent (Experimental): Hydrus Microstent implanted in the eye immediately following cataract surgery and placement of a monofocal intraocular lens (IOL)
  Interventions: Device: Hydrus Microstent; Procedure: Cataract surgery; Device: Monofocal IOL

INTERVENTIONS:
Device: Hydrus Microstent — Crescent-shaped nitinol device intended as a permanent implant to provide an outflow pathway for aqueous humor. The device is placed through the trabecular meshwork into Schlemm's canal immediately following placement of a monofocal IOL.
Procedure: Cataract surgery — Cataract surgery performed using standard anesthesia and phacoemulsification techniques
Device: Monofocal IOL — Commercially available monofocal intraocular lens as determined by the investigator

SUMMARY:
The purpose of this post-approval study is to evaluate the rate of Hydrus Microstent malposition and associated clinical sequelae occurring within 24 months post-operation. Qualified subjects will undergo uncomplicated cataract surgery with placement of a monofocal intraocular lens (IOL), followed by implantation of the Hydrus Microstent.

DETAILED DESCRIPTION:
Qualified subjects will attend a screening visit, a surgical visit (Day 0), and 8 scheduled postoperative visits at Day 1, Day 7, Month 1, Month 3, Month 6, Month 12, Month 18, and Month 24.

This study was initiated by Ivantis, Inc. Ivantis was acquired by Alcon Research, and Alcon assumed sponsorship of the study in November 2022.

ELIGIBILITY:
Inclusion Criteria:

* An operable, age-related cataract with best corrected visual acuity (BCVA) of 20/40 or worse;
* Diagnosis of primary open angle glaucoma treated with no more than 4 topical hypotensive medications;
* Optic nerve appearance characteristic of glaucoma;
* Medicated IOP less than or equal to 31 millimeters mercury (mmHg); Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Closed angle forms of glaucoma;
* Congenital or developmental glaucoma;
* Secondary glaucoma;
* Use of more than 4 ocular hypotensive medications;
* Previous argon laser trabeculoplasty, trabeculectomy, tube shunts, or any other prior filtration or cilioablative surgery;
* Prior surgery with implanted device or other surgery involving the trabecular meshwork or Schlemm's canal;
* Other protocol-defined exclusion criteria may apply.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 545 (Estimated)
Dates: Start 2020-08-25 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Rate of occurrence of clinically significant device malposition associated with clinical sequelae | Day 0 operative, up to Month 24 postoperative
  The position of the implant will be assessed visually intraoperatively and at each postoperative follow-up visit. Examples of clinically significant device malposition associated with clinical sequelae as listed in the protocol include secondary surgical intervention to modify device position or to remove the device (explantation), corneal endothelial touch by device, iris touch by the device associated with intraocular inflammation, pigment dispersion or other sequelae, central endothelial cell loss ≥30 percent, compromised corneal function, best-corrected visual acuity (BCVA) loss of 2 lines (10 letters) or more on the ETDRS chart, device obstruction requiring secondary surgical intervention, persistent anterior chamber inflammation with peripheral anterior synechiae, persistent anterior chamber inflammation without peripheral anterior synechiae, and chronic pain.

SECONDARY OUTCOMES:
Rate of occurrence of intraoperative ocular adverse events | Day 0 operative
  Intraoperative ocular adverse events as specified in the protocol include hyphema obscuring the surgeon's view, choroidal hemorrhage or effusion, choroidal detachment, significant iris injury or trauma, corneal abrasion, corneal edema, zonular dialysis, cyclodialysis, cyclodialysis cleft, iridodialysis, vitreous loss not associated with the cataract procedure, inadvertent perforation of the sclera, and Descemet's membrane detachment.
Rate of occurrence of sight threatening postoperative adverse events | Up to Month 24
  Sight threatening, post-operative adverse events as specified in the protocol include endophthalmitis, corneal decompensation, severe retinal detachment, severe choroidal hemorrhage, severe choroidal detachment, and aqueous misdirection.
Rate of occurrence of other postoperative ocular adverse events | Up to Month 24
  Other postoperative ocular adverse events as specified in the protocol include anterior uveitis/iritis, non-persistent & persistent, best corrected visual acuity (BCVA) loss of 2 lines or more, chronic pain, device migration, device obstruction, peripheral anterior synechiae (PAS), ocular secondary surgical interventions for intraocular pressure (IOP) or glaucoma management, hypotony at or after 1 month postop, hyphema, corneal opacification, corneal edema persisting or severe corneal edema, other retinal complications, elevated mean IOP >/=10 millimeters mercury (mmHg) vs screening, iris prolapse/wound incarceration, significant foreign body sensation at or after 3 months postop, surgical re-intervention, and worsening of visual field.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Project Lead, CDMA Surgical, Study Director — Alcon Research
Locations (22):
- United States (22):
  - Coastal Vision, Irvine, California
  - Sacramento Eye Consultants, Sacramento, California
  - Eye Center of Northern Colorado, Loveland, Colorado
  - Jones Eye Center PC, Sioux City, Iowa
  - Stiles Eyecare Excellence Cataracts and Glaucoma, Overland Park, Kansas
  - Visionary Eye Doctors, Rockville, Maryland
  - Fraser Eye Care Center, Fraser, Michigan
  - Twin Cities Eye Consultants, Coon Rapids, Minnesota
  - Midwest Vision Research Foundation, Chesterfield, Missouri
  - Moyes Eye Center, Kansas City, Missouri
  - Center for Sight, Las Vegas, Nevada
  - Carolina Eye Associates PA, Southern Pines, North Carolina
  - Cleveland Eye Clinic, Brecksville, Ohio
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Cincinnati Eye / Apex Eye, Mason, Ohio
  - Scott & Christie and Associates, PC, Cranberry Township, Pennsylvania
  - Texan Eye / Keystone Research, Austin, Texas
  - Glaucoma Associates Of Texas, Dallas, Texas
  - El Paso Eye Surgeons, El Paso, Texas
  - Texas Eye Research Center, Hurst, Texas
  - The Eye Institute of Utah, Salt Lake City, Utah
  - Eye Centers Of Racine And Kenosha, Kenosha, Wisconsin

IPD SHARING:
Plan to Share IPD: No